CLINICAL TRIAL: NCT02993471
Title: Evaluation of the Effect of Ixekizumab on the Pharmacokinetics of Cytochrome P450 Substrates in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of Ixekizumab in Participants With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16126; I1F-MC-RHBU (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2017-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Caffeine; Warfarin; Omeprazole; Dextromethorphan; Midazolam; ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Cocktail (Experimental): Drug cocktail (caffeine, warfarin [plus vitamin K], omeprazole, dextromethorphan, and midazolam) administered orally once in Period 1 (day 1).
  Interventions: Drug: Drug Cocktail
- Drug Cocktail + Ixekizumab (Experimental): Drug cocktail (caffeine, warfarin [plus vitamin K], omeprazole, dextromethorphan, and midazolam) administered orally twice in Period 2 (day 8 and day 85). Ixekizumab administered subcutaneously (SC) on multiple occasions in Period 2.
  Interventions: Drug: Drug Cocktail; Drug: Ixekizumab

INTERVENTIONS:
Drug: Drug Cocktail — Administered orally
  Other Names: Caffeine + Warfarin (plus vitamin K) + Omeprazole + Dextromethorphan + Midazolam
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Drug Cocktail + Ixekizumab

SUMMARY:
This study is known as a "drug interaction study." The purpose is to learn about how ixekizumab may affect the blood levels of a mixture of commonly used drugs (caffeine, omeprazole, warfarin, dextromethorphan, and midazolam) that are metabolized by cytochrome P450. Each participant will complete two study periods. Participants will take the mixture of commonly used drugs (plus vitamin K) by mouth on 3 occasions (prior to treatment with ixekizumab and after 1 and 12 weeks of treatment with ixekizumab). The study will last about 17 weeks, including follow-up. Screening must be completed prior to study start.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with chronic moderate or severe plaque psoriasis for at least 6 months who are candidates for systemic therapy or phototherapy
* Men and women of childbearing potential must agree to use a reliable method of birth control and men may not donate sperm for the duration of the study. Women must test negative for pregnancy at screening and agree not to become pregnant during the study and until the first normal period following the end of the study
* Have a body mass index (BMI) of 18.5 to 40.0 kilograms per square meter (kg/m²), inclusive, at screening
* Have greater than or equal to (≥) 10 percent body surface area (BSA) involvement at screening and first admission to the clinical research unit (CRU)
* Have both a Static Physicians Global Assessment (sPGA) score of ≥3 and Psoriasis Area Severity Index (PASI) score ≥12 at screening and first admission to the CRU

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type
* Pregnant or nursing (lactating women)
* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection
* Have major surgery within 8 weeks prior to first admission to the clinical research unit or during the study
* Have a history of lymphoproliferative disease, or signs or symptoms of lymphoproliferative disease, or have active or history of malignant disease, or have uncontrolled cerebrocardiovascular or neuropsychiatric disease
* Require treatment with the cocktail drugs or with inhibitors of cytochrome P450 (CYP) 3A, CYP2C9, CYP2D6, CYP2C19, CYP1A2, or with inducers of CYP3A or CYP1A2, or with rifampin (inducer of multiple CYPs) or with substrates of CYP3A, CYP2C9, CYP2D6, CYP2C19, or CYP1A2 with narrow therapeutic indices within 14 days prior to the first administration of the drug cocktail through the end of Week 12 assessments
* Have any known allergy or hypersensitivity to any component of the study cocktail or ixekizumab
* Have participated in any other study with ixekizumab, secukinumab or brodalumab, or have been prescribed ixekizumab or secukinumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Avail Clinical Research LLC, DeLand, Florida
  - High Point Clinical Trials Center, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: A Study of Ixekizumab in Participants with Plaque Psoriasis — https://www.lillytrialguide.com/en-US/studies/psoriasis/RHBU#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Multicenter, open-label, 2-period, fixed-sequence study.
Groups:
- Drug Cocktail /Drug Cocktail + Ixekizumab: Period 1: Participants received drug cocktail (100 mg Caffeine, 10 mg Warfarin [plus vitamin K], 20 mg Omeprazole, 30 mg Dextromethorphan, and 1 mg Midazolam) administered orally on Day 1. Participants resided at the Clinical Research Unit (CRU) until Day 2, and were discharged following collection of 24-hour pharmacokinetics (PK) samples for the determination of plasma concentrations of the cocktail drugs and metabolites.
  Period 2: Participants received a 160 mg dose of Ixekizumab during an outpatient visit on Day 1 (3 to 7 days after Day 5 of Period 1) and were admitted to the CRU on Day 7 (±2 days) to receive the drug cocktail on the morning of Day 8 (Week 1). Participants received single 80 mg doses of Ixekizumab at outpatient visits on Day 15 (Week 2), Day 29 (Week 4), Day 43 (Week 6), Day 57 (Week 8), and Day 71 (Week 10). Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg Ixekizumab and the drug cocktail on the following morning (Day 85; Week 12).
Period: Period 1 (Drug Cocktail)
Arm/Group | Drug Cocktail /Drug Cocktail + Ixekizumab
Started | 28
Received at Least 1 Dose of Study Drug | 28
Completed | 28
Not Completed | 0
Period: Period 2 (Drug Cocktail + Ixekizumab)
Arm/Group | Drug Cocktail /Drug Cocktail + Ixekizumab
Started | 28
Received at Least 1 Dose of Study Drug | 27
Completed | 26
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Overall Study: Participants received drug cocktail and drug cocktail + Ixekizumab.
Arm/Group | Overall Study
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Cytochrome P450 (CYP450) Substrate-Midazolam
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Cytochrome P450 (CYP450) Substrate (Midazolam)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 1 mg Midazolam: Participants received 1 mg of Midazolam on Day 1 of Period 1.
- 160 mg Ixekizumab + 1 mg Midazolam: Participants received 160 mg dose of Ixekizumab on Day 1 and 1 mg of Midazolam on Day 8 of Period 2.
- 80 mg Ixekizumab Q2W (Once Every Two Weeks) + 1 mg Midazolam: Participants received 80 mg of Ixekizumab on Day 15, Day 29, Day 43, Day 57, and Day 71. Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg of Ixekizumab and 1 mg of Midazolam on the following morning (Day 85; Week 12) during Period 2.
Arm/Group | 1 mg Midazolam | 160 mg Ixekizumab + 1 mg Midazolam | 80 mg Ixekizumab Q2W (Once Every Two Weeks) + 1 mg Midazolam
Number analyzed (Participants) | 27 | 26 | 25
nanogram per milliliter (ng/mL) | 4.56 (24) | 4.92 (24) | 4.83 (26)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of CYP450 Substrate-Midazolam
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Zero to Infinity (AUC[0-∞]) of CYP450 Substrate (Midazolam)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- 80 mg Ixekizumab Q2W + 1 mg Midazolam: Participants received 80 mg of Ixekizumab on Day 15, Day 29, Day 43, Day 57, and Day 71. Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg of Ixekizumab and 1 mg of Midazolam on the following morning (Day 85; Week 12) during Period 2.
Arm/Group | 1 mg Midazolam | 160 mg Ixekizumab + 1 mg Midazolam | 80 mg Ixekizumab Q2W + 1 mg Midazolam
Number analyzed (Participants) | 27 | 26 | 25
nanogram*hour per milliliter (ng*h/mL) | 16.6 (28) | 15.9 (27) | 15.4 (34)

3. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate-Warfarin
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate (Warfarin)
Time Frame: Predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 10 mg Warfarin: Participants received 10 mg of Warfarin on Day 1 of Period 1.
- 160 mg Ixekizumab + 10 mg Warfarin: Participants received 160 mg dose of Ixekizumab on Day 1 and 10 mg of Warfarin on Day 8 of Period 2.
- 80 mg Ixekizumab Q2W + 10 mg Warfarin: Participants received 80 mg of Ixekizumab on Day 15, Day 29, Day 43, Day 57, and Day 71. Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg of Ixekizumab and 10 mg of Warfarin on the following morning (Day 85; Week 12) during Period 2.
Arm/Group | 10 mg Warfarin | 160 mg Ixekizumab + 10 mg Warfarin | 80 mg Ixekizumab Q2W + 10 mg Warfarin
Number analyzed (Participants) | 27 | 26 | 25
ng/mL | 510 (26) | 525 (22) | 510 (23)

4. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of CYP450 Substrate-Warfarin
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Zero to Infinity (AUC[0-∞]) of CYP450 Substrate (Warfarin)
Time Frame: Predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, and 96 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 10 mg Warfarin | 160 mg Ixekizumab + 10 mg Warfarin | 80 mg Ixekizumab Q2W + 10 mg Warfarin
Number analyzed (Participants) | 27 | 26 | 25
ng*h/mL | 17600 (29) | 17700 (31) | 16200 (29)

5. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate-Dextromethorphan
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate (Dextromethorphan)
Time Frame: Predose, 1, 2, 4, 6, 8, 10, 24, 48, and 72 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 30 mg Dextromethorphan: Participants received 30 mg of Dextromethorphan on Day 1 of Period 1.
- 160 mg Ixekizumab + 30 mg Dextromethorphan: Participants received 160 mg dose of Ixekizumab on Day 1 and 30 mg of Dextromethorphan on Day 8 of Period 2.
- 80 mg Ixekizumab Q2W + 30 mg Dextromethorphan: Participants received 80 mg of Ixekizumab on Day 15, Day 29, Day 43, Day 57, and Day 71. Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg of Ixekizumab and 30 mg of Dextromethorphan on the following morning (Day 85; Week 12) during Period 2.
Arm/Group | 30 mg Dextromethorphan | 160 mg Ixekizumab + 30 mg Dextromethorphan | 80 mg Ixekizumab Q2W + 30 mg Dextromethorphan
Number analyzed (Participants) | 27 | 25 | 24
ng/mL | 0.691 (291) | 0.878 (202) | 0.658 (285)

6. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of CYP450 Substrate-Dextromethorphan
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Zero to Infinity (AUC[0-∞]) of CYP450 Substrate (Dextromethorphan)
Time Frame: Predose, 1, 2, 4, 6, 8, 10, 24, 48, and 72 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 30 mg Dextromethorphan | 160 mg Ixekizumab + 30 mg Dextromethorphan | 80 mg Ixekizumab Q2W + 30 mg Dextromethorphan
Number analyzed (Participants) | 25 | 24 | 23
ng*h/mL | 11.7 (254) | 12.6 (225) | 8.53 (273)

7. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate-Omeprazole and Its Metabolite 5-Hydroxyomeprazole
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate (Omeprazole and its metabolite 5-Hydroxyomeprazole)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 20 mg Omeprazole: Participants received 20 mg of Omeprazole on Day 1 of Period 1.
- 160 mg Ixekizumab + 20 mg Omeprazole: Participants received 160 mg dose of Ixekizumab on Day 1 and 20 mg of Omeprazole on Day 8 of Period 2.
- 80 mg Ixekizumab Q2W + 20 mg Omeprazole: Participants received 80 mg of Ixekizumab on Day 15, Day 29, Day 43, Day 57, and Day 71. Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg of Ixekizumab and 20 mg of Omeprazole on the following morning (Day 85; Week 12) during Period 2.
Arm/Group | 20 mg Omeprazole | 160 mg Ixekizumab + 20 mg Omeprazole | 80 mg Ixekizumab Q2W + 20 mg Omeprazole
Number analyzed (Participants) | 27 | 26 | 25
ng/mL
  Omeprazole | 333 (83) | 340 (74) | 368 (62)
  5-Hydroxyomeprazole | 148 (55) | 143 (57) | 137 (46)

8. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of CYP450 Substrate-Omeprazole and Its Metabolite 5-Hydroxyomeprazole
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Zero to Infinity (AUC[0-∞]) of CYP450 Substrate (Omeprazole and its metabolite 5-Hydroxyomeprazole)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 20 mg Omeprazole | 160 mg Ixekizumab + 20 mg Omeprazole | 80 mg Ixekizumab Q2W + 20 mg Omeprazole
Number analyzed (Participants) | 22 | 23 | 21
ng*h/mL
  Omeprazole | 1060 (104) | 829 (129) | 913 (107)
  5-Hydroxyomeprazole | 519 (28) | 475 (25) | 455 (24)

9. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate-Caffeine
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of CYP450 Substrate (Caffeine)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 100 mg Caffeine: Participants received 100 mg of Caffeine on Day 1 of Period 1.
- 160 mg Ixekizumab + 100 mg Caffeine: Participants received 160 mg dose of ixekizumab on Day 1 and 100 mg of Caffeine on Day 8 of Period 2.
- 80 mg Ixekizumab Q2W + 100 mg Caffeine: Participants received 80 mg of ixekizumab on Day 15, Day 29, Day 43, Day 57, and Day 71. Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg of ixekizumab and 100 mg of Caffeine on the following morning (Day 85; Week 12) during Period 2.
Arm/Group | 100 mg Caffeine | 160 mg Ixekizumab + 100 mg Caffeine | 80 mg Ixekizumab Q2W + 100 mg Caffeine
Number analyzed (Participants) | 18 | 21 | 13
ng/mL | 2230 (19) | 2220 (22) | 2240 (22)

10. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to 48 Hours (AUC[0-48h]) of CYP450 Substrate-Caffeine
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Zero to 48 hours (AUC[0-48h]) of CYP450 Substrate (Caffeine)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours postdose
Population: All enrolled participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 100 mg Caffeine | 160 mg Ixekizumab + 100 mg Caffeine | 80 mg Ixekizumab Q2W + 100 mg Caffeine
Number analyzed (Participants) | 13 | 19 | 11
ng*h/mL | 25000 (48) | 22400 (57) | 22400 (36)

ADVERSE EVENTS:
Time Frame: Up To 89 days
Description: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Drug Cocktail: Participants received drug cocktail (100 mg Caffeine, 10 mg Warfarin [plus vitamin K], 20 mg Omeprazole, 30 mg Dextromethorphan, and 1 mg Midazolam) administered orally on Day 1 of period 1.
- Drug Cocktail + Ixekizumab: Participants received a 160 mg dose of Ixekizumab during an outpatient visit on Day 1 (3 to 7 days after Day 5 of Period 1) and were admitted to the CRU on Day 7 (±2 days) to receive the drug cocktail on the morning of Day 8 (Week 1). Participants received single 80 mg doses of Ixekizumab at outpatient visits on Day 15 (Week 2), Day 29 (Week 4), Day 43 (Week 6), Day 57 (Week 8), and Day 71 (Week 10). Participants were admitted to the CRU on Day 84 (±2 days) and received 80 mg Ixekizumab and the drug cocktail on the following morning (Day 85; Week 12).
Arm/Group | Drug Cocktail | Drug Cocktail + Ixekizumab
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 1/28 | 7/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Cocktail (N=28) | Drug Cocktail + Ixekizumab (N=27)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT02993471/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT02993471/SAP_001.pdf